CLINICAL TRIAL: NCT07052578
Title: A Multicentre Observational Study on Treatment Patterns and ctDNA HRR Evaluation in Aggressive High-volume Metastatic Hormone-sensitive Prostate Cancer in Russian Federation
Brief Title: Aggressive Disease Treatment Patterns and CtDNA HRR evaluatiON in High-volume metastatiC hORmone-sensitive Prostate Cancer in Russian FeDeration
Acronym: CONCORD
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133HR00059
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
A multicentre observational study on treatment patterns and ctDNA HRR evaluation in aggressive high-volume metastatic hormone-sensitive prostate cancer in Russian Federation

DETAILED DESCRIPTION:
This is a multicentre observational study on treatment approaches, demographic and clinical characteristics and on HRRm evaluation in ctDNA in patients with high-aggressive high-volume mHSPC with known tumor HRRm status in Russian Federation. The study will sequentially include only those patients who have signed the informed consent form (ICF). No procedures will be applied to patients in addition to the routine clinical practice.

Study population will consist of patients with high-aggressive (Gleason 8-10) high-volume mHSPC with available medical history and known tumor HRRm status, which has been determined from a tumour sample obtained from the patient as part of routine practice. It is estimated that approximately 400 patients will be enrolled in about 30 sites. In this case, the ratio of patients with HRR gene mutations (HRRm) to patients with wild-type HRR genes (HRRwt) will be approximately 5:3 (250 HRRm and 150 HRRwt), so that both populations are represented in the study sample, including patients without mutations.

The study will include two visits carried out according to routine clinical practice. At baseline visit (visit 1) demographic and clinical characteristics and treatment approaches from the date of high-aggressive high-volume mPC diagnosis (date of first metastases verification) till enrollment will be collected based on the patient's medical records. In case of absence of data required to be collected by the protocol, additional data may be obtained during patient's interview directly and recorded in the source documents related to the visit. For ctDNA and ctDNA-based HRRm testing (by NGS) routinely collected blood samples will be used. Testing will be performed in central laboratories.

Visit 2 (final visit) will be conducted at the time of disease progression or after 12 (±3) months (whichever occurs first) to collect follow-up data on progression to mCRPC and subsequent treatment, if applicable. If the patient is unable to visit the study site (e.g. in case the patient is being treated and observed at the place of residence) the data collection of visits 2 could be carried out via telephone contact.

All study data will be entered into electronic case report form (eCRF). The study physician will be responsible for ensuring that all required data is collected and entered into the eCRF.

Overall expected duration of the study (from the first patient inclusion to the final database lock) is about 38 months, or until 400 eligible patients are included to the study and data on these patients are collected (including follow-up data), whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients aged ≥ 18 years old;
2. Signed ICF, including consent for blood samples ctDNA and ctDNA-based HRRm testing;
3. Metastatic hormone-sensitive prostate cancer (mHSPC) (de novo or progressed from earlier stages);
4. High-aggressive disease (Gleason 8-10);
5. High-volume disease (according to CHAARTED trial criteria: presence of 4 and more (≥4) bone metastases (including at least one (≥1) outside the vertebral column/pelvis) and/or 1 and more (≥1) visceral metastasis);
6. Availability of source medical documentation;
7. Known HRRm status based on tumour sample evaluation performed in routine practice.

Exclusion Criteria:

1. Participation in any interventional trial since the mPC diagnosis.
2. Progression to mCRPC.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to enroll approximately 400 patients with high-aggressive (Gleason 8-10) high-volume mHSPC (250 HRRm and 150 HRRwt) with available medical history and known HRRm status in about 30 sites in Russian Federation.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients received any ADT | 36 months
  Proportion of patients received any Androgen deprivation therapy
Proportion of patients received ADT by each type and by each drug | 36 months
  Proportion of patients received Androgen deprivation therapy by each type and by each drug
Proportion of patients received first generation antiandrogens | 36 months
  Proportion of patients received first generation antiandrogens
Proportion of patients received androgen receptor pathway inhibitors (ARPI) at mHSPC | 36 months
  Proportion of patients received androgen receptor pathway inhibitors (ARPI) at mHSPC overall and by each drug;
Duration of ARPI therapy | 36 months
  Duration (months) of androgen receptor pathway inhibitors (ARPI) therapy
Proportion of patients received any chemotherapy at mHSPC | 36 months
  Proportion of patients received any chemotherapy at metastatic hormone-sensitive prostate cancer
Duration of chemotherapy | 36 months
  Duration (months) of chemotherapy, No. of cycles of chemotherapy;
Proportion of patients received radiation therapy | 36 months
  Proportion of patients received radiation therapy (RT) overall and by each type (if applicable);
Proportion of patients with each radiation area | 36 months
  Proportion of patients with each radiation area (if applicable) (to be calculated in patients who received any RT);
Proportion of patients underwent surgery at mHSPC | 36 months
  Proportion of patients underwent surgery at Metastatic hormone-sensitive prostate cancer stage overall and by each type (if applicable);
Proportion of patients received triplet therapy at mHSPC | 36 months
  Proportion of patients received triplet therapy (ADT + ARPI + chemotherapy) at Metastatic hormone-sensitive prostate cancer overall and by each ARPI;
Time from mPC diagnosis to progression to mCRPC | 36 months
  Time from Metastatic prostate cancer diagnosis to progression to Metastatic castration-resistant prostate cancer (mCRPC) (calculated between the date of confirmed metastatic disease diagnosis and the date of progression to mCRPC) in the total sample and in different subgroups (HRRm/HRRwt, ctDNA+/ctDNA-, different therapeutical approaches);
Proportion of patients with each site of disease progression | 36 months
  Proportion of patients with each site of disease progression (metastases);
Testosterone level at the time of mCRPC | 36 months
  Testosterone level (nmol/l) at the time of castrate-resistant disease (mCRPC diagnosis);
Proportion of patients with presence of pathogenic mutations in HRR genes in ctDNA | 36 months
  Proportion of patients with presence of pathogenic mutations in Homologous recombination repair (HRR) genes detected in culating tumor DNA (ctDNA) by Next Generation Sequencing (NGS) overall and by each gene.

SECONDARY OUTCOMES:
Age at the diagnosis of high-aggressive high-volume mPC | 36 months
  Age at the diagnosis of high-aggressive high-volume Metastatic prostate cancer (mPC)
Proportion of patients of different races and ethnicities | 36 months
  Proportion of patients of different races and ethnicities overall and in subgroups HRRm/HRRwt;
Proportion of patients with presence of a family oncology history | 36 months
  Proportion of patients with presence of a family oncology history (first degree relatives) overall and by each disease, in the total sample and in subgroups HRRm/HRRwt;
Proportion of patients with a personal oncology history | 36 months
  Proportion of patients with a personal oncology history overall and by each disease, in the total sample and in subgroups HRRm/HRRwt;
Proportion of patients with each category by ECOG assessmen | 36 months
  Proportion of patients with each category by Eastern Cooperative Oncology Group (ECOG) assessment at the inclusion;
Proportion of patients with each type of mPC diagnosi | 36 months
  Proportion of patients with each type of Metastatic prostate cancer (mPC) diagnosis (de novo, metachronous);
Proportion of patients with each stage by TNM classification | 36 months
  Proportion of patients with each stage by TNM classification;
Proportion of patients with each histological type of tumor | 36 months
  Proportion of patients with each histological type of tumor (types of adenocarcinoma);
Proportion of patients with each category by Gleason scale | 36 months
  Proportion of patients with each category (8 (4+4), 8 (3+5), 8 (5+3), 9, 10)) by Gleason scale, in the total sample and in subgroups (de novo and in metachronous mPC, HRRm/HRRwt, ctDNA+/ctDNA-);
Time from initial diagnosis to mPC diagnosis | 36 months
  Time from initial diagnosis to mPC diagnosis (calculated for patients with metachronous disease, as a time period between the date of initial diagnosis of PC and the date of confirmed metastatic disease diagnosis);
Proportion of patients with each localization of metastases at the diagnosis of mPC | 36 months
  Proportion of patients with each localization of metastases at the diagnosis of mPC (confirmed metastatic disease), symptomatic or not;
PSA level at the diagnosis of mPC | 36 months
  PSA level at the diagnosis of mPC (confirmed metastatic disease);
Proportion of patients with each HRR mutation among all HRRm patient | 36 months
  Proportion of patients with each HRR mutation among all HRRm patients, in the total sample and in subgroups (de novo and in metachronous mPC, ctDNA+/ctDNA-);
Proportion of patients with each source of tumor sample | 36 months
  Proportion of patients with each source of tumor sample (primary tumor, metastases), which was used for the HRRm status determination in routine practice;
Proportion of patients with presence of ctDNA | 36 months
  Proportion of patients with presence of ctDNA, in the total sample and in subgroups (de novo and in metachronous mPC, HRRm/HRRwt);
ctDNA HRRm/HRRwt and tumor HRRm/HRRwt coincidence rate | 36 months
  ctDNA HRRm/HRRwt and tumor HRRm/HRRwt coincidence rate.

CONTACTS AND LOCATIONS:
Locations (16):
- Russia (16):
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Chelyabinsk
  - Research Site, Irkutsk
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Obninsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Sochi
  - Research Site, Tomsk
  - Research Site, Tver'
  - Research Site, Tyumen
  - Research Site, Ufa
  - Research Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Supporting Information: CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/